CLINICAL TRIAL: NCT02838407
Title: Identification and Characterization of Bacteria in the Lower Airways of Children Aged ≥ 6 Months to < 6 Years With Suspected Lower Respiratory Tract Infections (LRTI) in Spain.
Brief Title: Identification and Characterization of Bacteria in the Lungs of Children From 6 Months up to 6 Years Old, With Suspected Infection of the Lungs, in Spain.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 115813
Record Dates: First submitted 2016-07-08; First posted 2016-07-20 (Estimated); Results first posted 2019-10-04 (Actual); Last update posted 2019-10-04 (Actual); Status verified 2019-09

CONDITIONS: Infections, Streptococcal
Keywords: Chronic lower respiratory tract infection; Bonchoalveolar lavage; Nasopharyngeal swabs
MeSH Terms: conditions — Streptococcal Infections

ARMS (1):
- Total group (Other): All enrolled subjects, male or female aged between 6 months included and less than 6 years at the time of enrollment, who visited the hospital with suspected chronic lower respiratory tract infections (LRTIs) and who had an indication for bronchoalveolar lavage (BAL).
  Interventions: Other: BAL fluid sampling; Other: Nasopharyngeal swab sampling

INTERVENTIONS:
Other: BAL fluid sampling — Following routine BAL procedures at the hospital, collection of BAL fluid samples: at least 2 mL, at Day 0.
Other: Nasopharyngeal swab sampling — 1 swab, Day 0

SUMMARY:
The purpose of this study is to identify and characterise bacteria present in the lower airways of children with suspected chronic LRTIs and for whom bronchoalveolar lavage (BAL) is indicated by the clinician.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that parent(s)/ legally acceptable representatives (LAR[s]) can and will comply with the requirements of the protocol.
* A male or female subject aged ≥ 6 months to < 6 years at the time of enrolment.
* Subjects meet the case definition of suspected chronic LRTIs where BAL is indicated.
* Subject's parent(s)/ LAR(s) agree to the collection of a nasopharyngeal swab from the subject.
* Written informed consent obtained from the parent(s)/ LAR(s) of the subject.

Exclusion Criteria:

* Known cystic fibrosis, immunosuppression, or other severe immunodeficiencies such as agammaglobu-linaemia, T cell deficiency or Human Immunodeficiency Virus/ Acquired Immune Deficiency Syndrome, chemotherapy treatment, etc.
* Exacerbation of persistent respiratory symptoms (cough, wheezing, difficulty in breathing, etc.) in the previous 2 weeks.
* Antibiotic treatment in the 2 weeks prior to study entry.
* Concurrent participation in another study within 30 days prior to study entry or at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product (pharmaceutical product or device).
* Subjects having previously participated in this study.
* Child in care.

Ages: 6 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 197 (Actual)
Dates: Start 2013-09-23 (Actual); Primary Completion 2015-09-23 (Actual); Study Completion 2015-09-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (6):
- Spain (6):
  - GSK Investigational Site, Barakaldo (Vizcaya)
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Murcia (El Palmar)
  - GSK Investigational Site, Sabadell (Barcelona)
  - GSK Investigational Site, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Escribano Montaner A, Garcia de Lomas J, Villa Asensi JR, Asensio de la Cruz O, de la Serna Blazquez O, Santiago Burruchaga M, Mondejar Lopez P, Torrent Vernetta A, Feng Y, Van Dyke MK, Reyes J, Garcia-Corbeira P, Talarico CA; EPI-Strep-064 study group. Bacteria from bronchoalveolar lavage fluid from children with suspected chronic lower respiratory tract infection: results from a multi-center, cross-sectional study in Spain. Eur J Pediatr. 2018 Feb;177(2):181-192. doi: 10.1007/s00431-017-3044-3. Epub 2017 Dec 29. PMID 29285648

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Total Group
Started | 197
Completed | 197
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Total Group
Number analyzed (Participants) | 197
Age, Continuous [Mean (Standard Deviation); unit: Months] | 40.7 (18.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 95
  Male | 102

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Bacterial Aetiology, Assessed by Culture Growth, From Bronchoalveolar Lavage (BAL) Fluid Samples
Description: Bacterial aetiology was assessed by culture growth from BAL fluid sample for Steptococcus pneumoniae (S.p.), Haemophilus influenzae (H.i.) and Moraxella catarrhalis (M.c.) , through either qualitative or quantitative bacterial identification (B.I.). The categories assessed were: positive (Pos.), negative (Neg.) and Missing (Mis.). For quantitative bacterial identification, S.p., H.i. and M.c. were confirmed by bacterial identification load higher than (>) 10^4 colony forming units per milliliter (cfu/mL), if bacterial species were present alone, or >10^5 cfu/mL if present as co-infection.
  Note: For one subject who underwent BAL procedure, no BAL fluid was available for study analyses.
Time Frame: From Day 0 up to Year 2
Population: The analysis was performed on the According to protocol (ATP) cohort, which included all evaluable subjects, who complied with the protocol and with BAL fluid sampling results available.
Measure: Count of Participants; unit: Participants
Arm/Group | Total Group
Number analyzed (Participants) | 191
Participants
  Pos. qualitative B.I. for any of the 3 bacteria | 141
  Neg. qualitative B.I. for any of the 3 bacteria | 49
  Mis. qualitative B.I. for any of the 3 bacteria | 1
  Pos. qualitative B.I. for S. pneumoniae | 58
  Neg. qualitative B.I. for S. pneumoniae | 132
  Mis. qualitative B.I. for S. pneumoniae | 1
  Pos. qualitative B.I. for H. influenzae | 97
  Neg. qualitative B.I. for H. influenzae | 93
  Mis. qualitative B.I. for H. influenzae | 1
  Pos. qualitative B.I. for M. catarrhalis | 94
  Neg. qualitative B.I. for M. catarrhalis | 96
  Mis. qualitative B.I. for M. catarrhalis | 1
  Pos. qualitative B.I. for other bacteria | 12
  Neg. qualitative B.I. for other bacteria | 0
  Mis. qualitative B.I. for other bacteria | 179
  Pos. quantitative B.I. for any of the 3 bacteria | 42
  Neg. quantitative B.I. for any of the 3 bacteria | 148
  Mis. quantitative B.I. for any of the 3 bacteria | 1
  Pos. quantitative B.I. for S. pneumoniae | 20
  Neg. quantitative B.I. for S. pneumoniae | 170
  Mis. quantitative B.I. for S. pneumoniae | 1
  Pos. quantitative B.I. for H. influenzae | 17
  Neg. quantitative B.I. for H. influenzae | 173
  Mis. quantitative B.I. for H. influenzae | 1
  Pos. quantitative B.I. for M. catarrhalis | 12
  Neg. quantitative B.I. for M. catarrhalis | 178
  Mis. quantitative B.I. for M. catarrhalis | 1

2. Primary Outcome: Number of Subjects With Bacterial Aetiology Characteristics in BAL Fluid Samples
Description: S. pneumoniae (S.p.), H. influenzae (H.i.) and M. catarrhalis (M.c.) were confirmed by bacterial identification (B.I.) load higher than (>) 10^4 colony forming units per milliliter (cfu/mL), if bacterial species were present alone, or >10^5 cfu/mL if presented as co-infection. Analysis was also performed for other bacterial pathogens alone or as co-infection.
  Note: For one subject who underwent BAL procedure, no BAL fluid was available for study analyses
Time Frame: From Day 0 up to Year 2
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Total Group
Number analyzed (Participants) | 191
Participants
  S.p. alone (B.I. >10^4 cfu/mL) | 15
  H.i. alone (B.I. >10^4 cfu/mL) | 14
  M.c. alone (B.I. >10^4 cfu/mL) | 6
  Other bacterial pathogens - Any load | 12
  Other bacterial pathogens alone - Any load | 10
  S.p. and H.i. (B.I. >10^5 cfu/mL) | 1
  S.p. and M.c. (B.I. >10^5 cfu/mL) | 4
  H.i. and M.c. (B.I. >10^5 cfu/mL) | 2

3. Primary Outcome: Number of Subjects With Bacterial Identification >10^4 Cfu/mL in BAL Fluid Samples (S. Pneumoniae and H. Influenzae Results for the "Negative M. Catarrhalis" BAL Fluid Samples Results Category)
Description: S. pneumoniae, H. influenzae and M. catarrhalis were confirmed by bacterial identification load higher than (>) 10^4 colony forming units per milliliter (cfu/mL), if bacterial species were present alone. Bacterial load referred to Negative M. catarrhalis - Negative S. pneumoniae - Negative H. influenzae (N.M.c.-N.S.p.-N.H.i.), Negative M. catarrhalis - Negative S. pneumoniae - Positive H. influenzae (N.M.c.-N.S.p.-P.H.i.), Negative M. catarrhalis - Positive S. pneumoniae - Negative H. influenzae (N.M.c.-P.S.p.-N.H.i.), Negative M. catarrhalis - Positive S. pneumoniae - Positive H. influenzae (N.M.c.-P.S.p.-P..H.i.).
  Notes: bacterial identification for the N.M.c.-P.S.p.-P.H.i. category was confirmed as a co-infection with a bacterial load >10^5 cfu/mL. For one subject who underwent BAL procedure, no BAL fluid was available for study analyses.
Time Frame: From Day 0 up to Year 2
Population: The analysis was performed on the According to protocol (ATP) cohort, which included all evaluable subjects, who complied with the protocol and with negative M.catarrhalis BAL Fluid samples results available.
Measure: Count of Participants; unit: Participants
Arm/Group | Total Group
Number analyzed (Participants) | 178
Participants
  N.M.c.-N.S.p.-N.H.i. | 148
  N.M.c.-N.S.p.-P.H.i. | 14
  N.M.c.-P.S.p.-N.H.i. | 15
  N.M.c.-P.S.p.-P.H.i. | 1

4. Primary Outcome: Number of Subjects With Bacterial Identification >10^4 Cfu/mL in BAL Fluid Samples (S. Pneumoniae and H. Influenzae Results for the "Positive M. Catarrhalis" BAL Fluid Samples Results Category)
Description: S. pneumoniae, H. influenzae and M. catarrhalis were confirmed by bacterial identification load higher than (>) 10^4 colony forming units per milliliter (cfu/mL), if bacterial species were present alone and by bacterial load >10^5 cfu/mL if presented as co-infection.
  Categories referred to Positive M. catarrhalis -Negative S. pneumoniae - Negative H. influenzae (P.M.c.-N.S.p.-N.H.i.), Positive M. catarrhalis -Negative S. pneumoniae - Positive H. influenzae (P.M.c.-N.S.p.-P.H.i.), Positive M. catarrhalis - Positive S. pneumoniae - Negative H. influenzae (P.M.c.-P.S.p.-N.H.i.), Positive M. catarrhalis - Positive S. pneumoniae - Positive H. influenzae (P.M.c.-P.S.p.-P.H.i.). Notes: bacterial identification for the P.M.c.-N.S.p.-P.H.i., P.M.c.-P.S.p.-N.H.i. and P.M.c.-P.S.p.-P.H.i. categories was confirmed by a bacterial identification >10^5 cfu/mL. For one subject who underwent BAL procedure, no BAL fluid was available for study analyses
Time Frame: From Day 0 up to Year 2
Population: The analysis was performed on the According to protocol (ATP) cohort, which included all evaluable subjects, who complied with the protocol and with positive M.catarrhalis BAL Fluid samples results available.
Measure: Count of Participants; unit: Participants
Arm/Group | Total Group
Number analyzed (Participants) | 12
Participants
  P.M.c.-N.S.p.-N.H.i. | 6
  P.M.c.-N.S.p.-P.H.i. | 2
  P.M.c.-P.S.p.-N.H.i. | 4
  P.M.c.-P.S.p.-P.H.i. | 0

5. Secondary Outcome: Number of Subjects With Bacterial Colonization, Assessed by Culture Growth, From Nasopharyngeal Swab Samples
Description: Bacterial colonization was assessed by culture growth from nasopharyngeal swab samples for S. pneumoniae, H. influenzae and M. catarrhalis, through either qualitative or quantitative bacterial identification (B.I.). The categories assessed were: positive (Pos.) and negative (Neg.).
Time Frame: From Day 0 up to Year 2
Population: The analysis was performed on the According to protocol (ATP) cohort, which included all evaluable subjects, who complied with the protocol and with nasopharyngeal swab sampling results available.
Measure: Count of Participants; unit: Participants
Arm/Group | Total Group
Number analyzed (Participants) | 191
Participants
  Pos. qualitative B.I. for any of the 3 bacteria | 154
  Neg. qualitative B.I. for any of the 3 bacteria | 37
  Pos. qualitative B.I. for S. pneumoniae | 99
  Neg. qualitative B.I. for S. pneumoniae | 92
  Pos. qualitative B.I. for H. influenzae | 89
  Neg. qualitative B.I. for H. influenzae | 102
  Pos. qualitative B.I. for M. catarrhalis | 107
  Neg. qualitative B.I. for M. catarrhalis | 84
  Pos. quantitative B.I. for any of the 3 bacteria | 37
  Neg. quantitative B.I. for any of the 3 bacteria | 154
  Pos. quantitative B.I. for S. pneumoniae | 24
  Neg. quantitative B.I. for S. pneumoniae | 167
  Pos. quantitative B.I. for H. influenzae | 7
  Neg. quantitative B.I. for H. influenzae | 184
  Pos. quantitative B.I. for M. catarrhalis | 10
  Neg. quantitative B.I. for M. catarrhalis | 181

6. Secondary Outcome: Bacterial Load Detected (log10 Transformation) by Quantitative Culture Growth, From BAL Fluid Samples
Description: Bacterial load was detected by quantitative culture growth from BAL fluid samples for S. pneumoniae, H. influenzae and M. catarrhalis and expressed in colony-forming unit/ milliliter (cfu/mL). Quantitative bacterial identification was used to indicate the presence of bacterial pathogen load >10^4 cfu/mL if present alone or > 10^5 cfu/mL if present as co-infection. Note: For one subject who underwent BAL procedure, no BAL fluid was available for study analyses.
Time Frame: From Day 0 up to Year 2
Population: The analysis was performed on the According to protocol (ATP) cohort, which included all evaluable subjects, who complied with the protocol and with BAL fluid sampling results available for the outcome measure.
Measure: Mean (Standard Deviation); unit: cfu/mL
Arm/Group | Total Group
Number analyzed (Participants) | 97
cfu/mL
  S. pneumoniae Bacterial load: number analyzed (Participants) | 58
  S. pneumoniae Bacterial load | 4.28 (1.04)
  H. influenzae Bacterial load | 3.81 (1.11)
  M. catarrhalis Bacterial load: number analyzed (Participants) | 94
  M. catarrhalis Bacterial load | 3.54 (1.01)

7. Secondary Outcome: Bacterial Load Detected (log10 Transformation) by Quantitative Molecular Techniques (Polymerase Chain Reaction) From BAL Fluid Samples
Description: Bacterial load was detected by quantitative molecular techniques (PCR) from BAL fluid samples for S. pneumoniae, H. influenzae and M. catarrhalis and expressed in colony-forming unit/milliliter (cfu/mL). Quantitative bacterial identification was used to indicate the presence of bacterial pathogen load >10^4 cfu/mL if present alone or > 10^5 cfu/mL if present as co-infection.
  Note: For one subject who underwent BAL procedure, no BAL fluid was available for study analyses.
Time Frame: From Day 0 up to Year 2
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: cfu/mL
Arm/Group | Total Group
Number analyzed (Participants) | 138
cfu/mL
  S. pneumoniae Bacterial load: number analyzed (Participants) | 105
  S. pneumoniae Bacterial load | 4.06 (1.27)
  H. influenzae Bacterial load | 4.31 (1.32)
  M. catarrhalis Bacterial load: number analyzed (Participants) | 128
  M. catarrhalis Bacterial load | 3.92 (1.29)

8. Secondary Outcome: Number of Subjects With Other Bacterial Pathogens Detected by Qualitative Culture, From BAL Fluid Samples
Description: Bacterial pathogens were detected by qualitative culture from BAL fluid samples and included:
  Staphylococcus aureus, Pseudomonas aeruginosa, Stenotrophomonas maltophilia and Pseudomonas putida.
  Note: For one subject who underwent BAL procedure, no BAL fluid was available for study analyses.
Time Frame: From Day 0 up to Year 2
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Total Group
Number analyzed (Participants) | 191
Participants
  Staphylococcus aureus (Growth) | 1
  Pseudomonas aeruginosa (Growth) | 5
  Stenotrophomonas maltophilia (Growth) | 4
  Pseudomonas putida (Growth) | 2

9. Secondary Outcome: Bacterial Load Detected (log10 Transformation) by Quantitative Culture From Nasopharyngeal Swab Samples
Description: Bacterial load was detected by quantitative culture from nasopharyngeal swab samples for S. pneumoniae, H. influenzae and M. catarrhalis and expressed in colony-forming unit/ milliliter (cfu/mL). Quantitative bacterial identification was used to indicate the presence of bacterial pathogen load >10^4 cfu/mL if present alone or > 10^5 cfu/mL if present as co-infection.
Time Frame: From Day 0 up to Year 2
Population: The analysis was performed on the According to protocol (ATP) cohort, which included all evaluable subjects, who complied with the protocol and with nasopharyngeal swab sampling results available for the outcome measure.
Measure: Mean (Standard Deviation); unit: cfu/mL
Arm/Group | Total Group
Number analyzed (Participants) | 107
cfu/mL
  S. pneumoniae Bacterial load: number analyzed (Participants) | 99
  S. pneumoniae Bacterial load | 3.99 (1.15)
  H. influenzae Bacterial load: number analyzed (Participants) | 89
  H. influenzae Bacterial load | 3.61 (0.88)
  M. catarrhalis Bacterial load | 3.36 (1.05)

10. Secondary Outcome: Bacterial Load Detected (log10 Transformation) by Molecular Techniques (PCR) From Nasopharyngeal Swab Samples
Description: Bacterial load was detected by quantitative molecular techniques from nasopharyngeal swab samples for S. pneumoniae, H. influenzae and M. catarrhalis and expressed in colony-forming unit/milliliter (cfu/mL). Quantitative bacterial identification was used to indicate the presence of bacterial pathogen load >10^4 cfu/mL if present alone or > 10^5 cfu/mL if present as co-infection.
Time Frame: From Day 0 and up to Year 2
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: cfu/mL
Arm/Group | Total Group
Number analyzed (Participants) | 133
cfu/mL
  S. pneumoniae Bacterial load: number analyzed (Participants) | 122
  S. pneumoniae Bacterial load | 4.39 (1.13)
  H. influenzae Bacterial load: number analyzed (Participants) | 122
  H. influenzae Bacterial load | 4.16 (1.17)
  M. catarrhalis Bacterial load | 4.05 (1.24)

11. Secondary Outcome: Number of Subjects With Other Bacterial Pathogens Detected by Qualitative Culture From Nasopharyngeal Swab Samples
Description: Bacterial pathogens were detected by qualitative culture from nasopharyngeal swab samples and included: Staphylococcus aureus and Stenotrophomonas maltophilia
Time Frame: From Day 0 and up to Year 2
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Total Group
Number analyzed (Participants) | 191
Participants
  Staphylococcus aureus (Growth) | 6
  Stenotrophomonas maltophilia (Growth) | 1

12. Secondary Outcome: Number of Qualitative Positive Unique Isolates of Subjects With S. Pneumoniae Serogroups and Serotypes in BAL Fluid Samples
Description: Two isolates of S.p., H.i. and M.c. were selected per specimen type per subjects. For analyses, the 2 isolates were compared to determine if they were clones vs. different ("unique") pathogen. Isolates were considered "unique" based on the comparison of serotype and antibiotic susceptibility (AS) profile for S.p. and H.i. and on the AS profile alone for M.c.. If the 2 isolates had different serotypes, or the same serotype but a different AS profile, then the 2 isolates were considered "unique", and both isolates were retained in the analyses. S.p. serogoups and serotypes isolates included: 3, 6B, 7C, 10A, 11A, 11D, 12F, 14, 15B, 16F, 18C, 18F, 19A, 19F, 21, 22F, 23A, 23B, 31, 35F, 42, 48, NT (not typeable), Synflorix serotypes (1, 4, 5, 6B, 7F, 9V, 14, 18C, 19A, 19F, 23F) and Pneumococcal conjugate vaccine (PCV) 13 serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, 23F). Note: For one subject who underwent BAL procedure, no BALF was available for study analyses.
Time Frame: From Day 0 to Year 2
Population: The analysis was performed on the According to protocol (ATP) cohort, which included all evaluable unique isolates of subjects for S. pneumoniae, who complied with the protocol and with BAL fluid sampling results available.
Measure: Number; unit: unique isolates of subjects
Arm/Group | Total Group
Number analyzed (Participants) | 65
unique isolates of subjects
  3 | 2
  6B | 4
  7C | 1
  10A | 3
  11A | 1
  11D | 4
  12F | 1
  14 | 3
  15B | 1
  16F | 2
  18C | 1
  18F | 10
  19A | 3
  19F | 4
  21 | 4
  22F | 2
  23A | 4
  23B | 1
  31 | 4
  35F | 3
  42 | 2
  48 | 1
  NT | 4
  Synflorix serotypes | 15
  PCV13 serotypes | 17

13. Secondary Outcome: Number of Qualitative Positive Unique Isolates of Subjects With H. Influenzae Typing Results From BAL Fluid Samples
Description: The H. influenzae typing results included "f" and "NT" (not typeable). Unique isolate definition: 2 isolates of S.p., H.i. and M.c. were selected per specimen type per subjects. For analyses, the 2 isolates were compared to determine if they were clones vs. different ("unique") pathogen. Isolates were considered "unique" based on the comparison of serotype and antibiotic susceptibility (AS) profile for S.p. and H.i. and on the AS profile alone for M.c.. If the 2 isolates had different serotypes, or the same serotype but a different AS profile, then the 2 isolates were considered "unique", and both isolates were retained in the analyses.
  Note: For one subject who underwent BAL procedure, no BALF was available for study analyses.
Time Frame: From Day 0 to Year 2
Population: The analysis was performed on the According to protocol (ATP) cohort, which included all evaluable unique isolates of subjects for H. influenzae, who complied with the protocol and with BAL fluid sampling results available.
Measure: Number; unit: unique isolates of subjects
Arm/Group | Total Group
Number analyzed (Participants) | 98
unique isolates of subjects
  f | 3
  NT | 95

14. Secondary Outcome: Number of Qualitative Positive Unique Isolates of Subjects With S. Pneumoniae Serogroups and Serotypes From Nasopharyngeal Swab Samples
Description: S. pneumoniae serogoups and serotypes included: 3, 6A, 6B, 7C, 9N, 10A, 11A, 11D, 12B, 12F, 14, 16F, 18C, 18F, 19A, 19C, 19F, 21, 23A, 23B, 31, 35A, 35F, 42, 48, NT (not typeable), Synflorix serotypes (1, 4, 5, 6B, 7F, 9V, 14, 18C, 19A, 19F, 23F) and Pneumococcal conjugate vaccine (PCV) 13 serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, 23F).
  Unique isolate definition: 2 isolates of S.p., H.i. and M.c. were selected per specimen type per subjects. For analyses, the 2 isolates were compared to determine if they were clones vs. different ("unique") pathogen. Isolates were considered "unique" based on the comparison of serotype and antibiotic susceptibility (AS) profile for S.p. and H.i. and on the AS profile alone for M.c.. If the 2 isolates had different serotypes, or the same serotype but a different AS profile, then the 2 isolates were considered "unique", and both isolates were retained in the analyses.
Time Frame: From Day 0 to Year 2
Population: The analysis was performed on the According to protocol (ATP) cohort, which included all evaluable unique isolates of subjects for S. pneumoniae, who complied with the protocol and with nasopharyngeal swab sampling results available.
Measure: Number; unit: unique isolates of subjects
Arm/Group | Total Group
Number analyzed (Participants) | 105
unique isolates of subjects
  3 | 2
  6A | 1
  6B | 6
  7C | 2
  9N | 1
  10A | 5
  11A | 1
  11D | 5
  12B | 1
  12F | 3
  14 | 2
  16F | 3
  18C | 1
  18F | 14
  19A | 6
  19C | 1
  19F | 9
  21 | 7
  23A | 5
  23B | 2
  31 | 3
  35A | 1
  35F | 3
  42 | 6
  48 | 4
  NT | 11
  Synflorix serotypes | 24
  PCV13 serotypes | 27

15. Secondary Outcome: Number of Qualitative Positive Unique Isolates of Subjects With H. Influenzae Typing Results From Nasopharyngeal Swab Samples
Description: The H. influenzae typing results include "f " and "NT" (not typeable). Unique isolate definition: 2 isolates of S.p., H.i. and M.c. were selected per specimen type per subjects. For analyses, the 2 isolates were compared to determine if they were clones vs. different ("unique") pathogen. Isolates were considered "unique" based on the comparison of serotype and antibiotic susceptibility (AS) profile for S.p. and H.i. and on the AS profile alone for M.c.. If the 2 isolates had different serotypes, or the same serotype but a different AS profile, then the 2 isolates were considered "unique", and both isolates were retained in the analyses.
Time Frame: From Day 0 to Year 2
Population: The analysis was performed on the According to protocol (ATP) cohort, which included all evaluable unique isolates of subjects for H. influenzae, who complied with the protocol and with nasopharyngeal swab sampling results available.
Measure: Number; unit: unique isolates of subjects
Arm/Group | Total Group
Number analyzed (Participants) | 92
unique isolates of subjects
  f | 4
  NT | 88

16. Secondary Outcome: Number of S. Pneumoniae Unique Isolates With Antimicrobial Susceptibility Response, Among Qualitative Positive Subjects
Description: Antibiotic response of S.pneumoniae was susceptible (Sus), or intermediate (Int), or resistant (Res)(following Clinical and Laboratory Standards Institute [CLSI] guidelines [CLSI, 2015]) towards the tested antibiotics which included: Penicilin, Amoxicillin/Clavulanate, Erythromycin, Azithromycin, Tetracycline, Levofloxacin, Trimethoprim/Sulfamethoxazole.
  Samples assessed were BAL fluid (BALF) samples and Nasopharyngeal swab (NPS) samples.
  For the "Unique isolate definition", please refer to the previous outcome description.
  Note: For one subject who underwent BAL procedure, no BAL fluid was available for study analyses.
Time Frame: From Day 0 to Year 2
Population: The analysis was performed on the S. pneumoniae unique isolates from qualitative positive subjects who were included in the ATP cohort.
Measure: Number; unit: unique isolates of subjects
Arm/Group | Total Group
Number analyzed (Participants) | 105
unique isolates of subjects
  Sus. Penicilin (BALF): number analyzed (Participants) | 65
  Sus. Penicilin (BALF) | 36
  Int. Penicilin (BALF): number analyzed (Participants) | 65
  Int. Penicilin (BALF) | 13
  Res. Penicilin (BALF): number analyzed (Participants) | 65
  Res. Penicilin (BALF) | 16
  Sus. Penicilin (NPS) | 55
  Int. Penicilin (NPS) | 27
  Res. Penicilin (NPS) | 23
  Sus. Amoxicillin/ Clavulanate (BALF): number analyzed (Participants) | 65
  Sus. Amoxicillin/ Clavulanate (BALF) | 50
  Int. Amoxicillin/ Clavulanate (BALF): number analyzed (Participants) | 65
  Int. Amoxicillin/ Clavulanate (BALF) | 7
  Res. Amoxicillin/ Clavulanate (BALF): number analyzed (Participants) | 65
  Res. Amoxicillin/ Clavulanate (BALF) | 8
  Sus. Amoxicillin/ Clavulanate (NPS) | 86
  Int. Amoxicillin/ Clavulanate (NPS) | 10
  Res. Amoxicillin/ Clavulanate (NPS) | 9
  Sus. Erythromycin (BALF): number analyzed (Participants) | 65
  Sus. Erythromycin (BALF) | 43
  Int. Erythromycin (BALF): number analyzed (Participants) | 65
  Int. Erythromycin (BALF) | 1
  Res. Erythromycin (BALF): number analyzed (Participants) | 65
  Res. Erythromycin (BALF) | 21
  Sus. Erythromycin (NPS) | 55
  Int. Erythromycin (NPS) | 1
  Res. Erythromycin (NPS) | 49
  Sus. Azithromycin (BALF): number analyzed (Participants) | 65
  Sus. Azithromycin (BALF) | 41
  Int. Azithromycin (BALF): number analyzed (Participants) | 65
  Int. Azithromycin (BALF) | 3
  Res. Azithromycin (BALF): number analyzed (Participants) | 65
  Res. Azithromycin (BALF) | 21
  Sus. Azithromycin (NPS) | 57
  Int. Azithromycin (NPS) | 4
  Res. Azithromycin (NPS) | 44
  Sus. Tetracycline (BALF): number analyzed (Participants) | 65
  Sus. Tetracycline (BALF) | 51
  Int. Tetracycline (BALF): number analyzed (Participants) | 65
  Int. Tetracycline (BALF) | 14
  Res. Tetracycline (BALF): number analyzed (Participants) | 65
  Res. Tetracycline (BALF) | 0
  Sus. Tetracycline (NPS) | 71
  Int. Tetracycline (NPS) | 3
  Res. Tetracycline (NPS) | 31
  Sus. Levofloxacin (BALF): number analyzed (Participants) | 65
  Sus. Levofloxacin (BALF) | 65
  Int. Levofloxacin (BALF): number analyzed (Participants) | 65
  Int. Levofloxacin (BALF) | 0
  Res. Levofloxacin (BALF): number analyzed (Participants) | 65
  Res. Levofloxacin (BALF) | 0
  Sus. Levofloxacin (NPS) | 103
  Int. Levofloxacin (NPS) | 0
  Res. Levofloxacin (NPS) | 2
  Sus. Trimethoprim/Sulfamethoxazole (BALF): number analyzed (Participants) | 65
  Sus. Trimethoprim/Sulfamethoxazole (BALF) | 24
  Int. Trimethoprim/Sulfamethoxazole (BALF): number analyzed (Participants) | 65
  Int. Trimethoprim/Sulfamethoxazole (BALF) | 13
  Res. Trimethoprim/Sulfamethoxazole (BALF): number analyzed (Participants) | 65
  Res. Trimethoprim/Sulfamethoxazole (BALF) | 28
  Sus. Trimethoprim/Sulfamethoxazole (NPS) | 52
  Int. Trimethoprim/Sulfamethoxazole (NPS) | 13
  Res. Trimethoprim/Sulfamethoxazole (NPS) | 40

17. Secondary Outcome: Number of H. Influenzae Unique Isolates With Antimicrobial Susceptibility Response, Among Qualitative Positive Subjects
Description: Antibiotic response of H.ifluenzae was susceptible (Sus), or intermediate (Int), or resistant (Res)(following Clinical and Laboratory Standards Institute [CLSI] guidelines [CLSI, 2015]) towards the tested antibiotics which included: Amoxicillin/Clavulanate, Azithromycin, Tetracycline, Levofloxacin, Trimethoprim/Sulfamethoxazole.
  Samples assessed were BAL fluid (BALF) samples and Nasopharyngeal swab (NPS) samples.
  For the "Unique isolate definition", please refer to the previous outcomes description.
  Note: For one subject who underwent BAL procedure, no BAL fluid was available for study analyses.
Time Frame: From Day 0 to Year 2
Population: The analysis was performed on the H. influenzae unique isolates from qualitative positive subjects who were included in the ATP cohort.
Measure: Number; unit: unique isolates of subjects
Arm/Group | Total Group
Number analyzed (Participants) | 98
unique isolates of subjects
  Sus. Amoxicillin/ Clavulanate (BALF) | 91
  Int. Amoxicillin/ Clavulanate (BALF) | 0
  Res. Amoxicillin/ Clavulanate (BALF) | 7
  Sus. Amoxicillin/ Clavulanate (NPS): number analyzed (Participants) | 92
  Sus. Amoxicillin/ Clavulanate (NPS) | 91
  Int. Amoxicillin/ Clavulanate (NPS): number analyzed (Participants) | 92
  Int. Amoxicillin/ Clavulanate (NPS) | 0
  Res. Amoxicillin/ Clavulanate (NPS): number analyzed (Participants) | 92
  Res. Amoxicillin/ Clavulanate (NPS) | 1
  Sus. Azithromycin (BALF) | 95
  Int. Azithromycin (BALF) | 0
  Res. Azithromycin (BALF) | 3
  Sus. Azithromycin (NPS): number analyzed (Participants) | 92
  Sus. Azithromycin (NPS) | 89
  Int. Azithromycin (NPS): number analyzed (Participants) | 92
  Int. Azithromycin (NPS) | 0
  Res. Azithromycin (NPS): number analyzed (Participants) | 92
  Res. Azithromycin (NPS) | 3
  Sus. Tetracycline (BALF) | 98
  Int. Tetracycline (BALF) | 0
  Res. Tetracycline (BALF) | 0
  Sus. Tetracycline (NPS): number analyzed (Participants) | 92
  Sus. Tetracycline (NPS) | 92
  Int. Tetracycline (NPS): number analyzed (Participants) | 92
  Int. Tetracycline (NPS) | 0
  Res. Tetracycline (NPS): number analyzed (Participants) | 92
  Res. Tetracycline (NPS) | 0
  Sus. Levofloxacin (BALF) | 98
  Int. Levofloxacin (BALF) | 0
  Res. Levofloxacin (BALF) | 0
  Sus. Levofloxacin (NPS): number analyzed (Participants) | 92
  Sus. Levofloxacin (NPS) | 92
  Int. Levofloxacin (NPS): number analyzed (Participants) | 92
  Int. Levofloxacin (NPS) | 0
  Res. Levofloxacin (NPS): number analyzed (Participants) | 92
  Res. Levofloxacin (NPS) | 0
  Sus. Trimethoprim/Sulfamethoxazole (BALF) | 51
  Int. Trimethoprim/Sulfamethoxazole (BALF) | 16
  Res. Trimethoprim/Sulfamethoxazole (BALF) | 31
  Sus. Trimethoprim/Sulfamethoxazole (NPS): number analyzed (Participants) | 92
  Sus. Trimethoprim/Sulfamethoxazole (NPS) | 49
  Int. Trimethoprim/Sulfamethoxazole (NPS): number analyzed (Participants) | 92
  Int. Trimethoprim/Sulfamethoxazole (NPS) | 18
  Res. Trimethoprim/Sulfamethoxazole (NPS): number analyzed (Participants) | 92
  Res. Trimethoprim/Sulfamethoxazole (NPS) | 25

18. Secondary Outcome: Descriptive Statistics of the Antimicrobial Susceptibility Response of H. Influenzae for Unique Isolates Among Qualitative Positive Subjects, for Penicilin and Erythromycin
Description: Antibiotic response of H. influenzae was tested against antibiotics which included: Penicilin and Erythromycin (following Clinical and Laboratory Standards Institute [CLSI] guidelines [CLSI, 2015]).
  Samples assessed were BAL fluid (BALF) samples and Nasopharyngeal swab (NPS) samples.
  Unique isolate definition: 2 isolates of S.p., H.i. and M.c. were selected per specimen type per subjects. For analyses, the 2 isolates were compared to determine if they were clones vs. different ("unique") pathogen. Isolates were considered "unique" based on the comparison of serotype and antibiotic susceptibility (AS) profile for S.p. and H.i. and on the AS profile alone for M.c.. If the 2 isolates had different serotypes, or the same serotype but a different AS profile, then the 2 isolates were considered "unique", and both isolates were retained in the analyses.
  Note: For one subject who underwent BAL procedure, no BAL fluid was available for study analyses.
Time Frame: From Day 0 to Year 2
Population: as for outcome 17
Measure: Median (Full Range); unit: unique isolates of subjects
Arm/Group | Total Group
Number analyzed (Participants) | 98
unique isolates of subjects
  Penicilin (BALF) | 0.5 [0.13 to 16.00]
  Penicilin (NPS): number analyzed (Participants) | 92
  Penicilin (NPS) | 0.5 [0.13 to 16.00]
  Erythromycin (BALF) | 4 [1.00 to 16.00]
  Erythromycin (NPS): number analyzed (Participants) | 92
  Erythromycin (NPS) | 4.00 [0.25 to 16.00]

19. Secondary Outcome: Number of M. Catarrhalis Unique Isolates With Antimicrobial Susceptibility Response, Among Qualitative Positive Subjects
Description: Antibiotic response of M. catarrhalis was susceptible (Sus), or intermediate (Int), or resistant (Res)(following Clinical and Laboratory Standards Institute [CLSI] guidelines [CLSI, 2015]) towards the tested antibiotics which included: Amoxicillin/Clavulanate, Erythromycin, Azithromycin, Tetracycline, Levofloxacin, Trimethoprim/Sulfamethoxazole.
  Samples assessed were BAL fluid (BALF) samples and Nasopharyngeal swab (NPS) samples.
  For the "Unique isolate definition", please refer to the previous outcome description.
  Note: For one subject who underwent BAL procedure, no BAL fluid was available for study analyses.
Time Frame: From Day 0 to Year 2
Population: The analysis was performed on the M. catarrhalis unique isolates from qualitative positive subjects who were included in the ATP cohort.
Measure: Number; unit: unique isolates of subjects
Arm/Group | Total Group
Number analyzed (Participants) | 110
unique isolates of subjects
  Sus. Amoxicillin/Clavulanate (BALF): number analyzed (Participants) | 98
  Sus. Amoxicillin/Clavulanate (BALF) | 95
  Int. Amoxicillin/Clavulanate (BALF): number analyzed (Participants) | 98
  Int. Amoxicillin/Clavulanate (BALF) | 0
  Res. Amoxicillin/Clavulanate (BALF): number analyzed (Participants) | 98
  Res. Amoxicillin/Clavulanate (BALF) | 3
  Sus. Amoxicillin/Clavulanate (NPS) | 105
  Int. Amoxicillin/Clavulanate (NPS) | 0
  Res. Amoxicillin/Clavulanate (NPS) | 5
  Sus. Erythromycin (BALF): number analyzed (Participants) | 98
  Sus. Erythromycin (BALF) | 90
  Int. Erythromycin (BALF): number analyzed (Participants) | 98
  Int. Erythromycin (BALF) | 0
  Res. Erythromycin (BALF): number analyzed (Participants) | 98
  Res. Erythromycin (BALF) | 8
  Sus. Erythromycin (NPS) | 106
  Int. Erythromycin (NPS) | 0
  Res. Erythromycin (NPS) | 4
  Sus. Azithromycin (BALF): number analyzed (Participants) | 98
  Sus. Azithromycin (BALF) | 84
  Int. Azithromycin (BALF): number analyzed (Participants) | 98
  Int. Azithromycin (BALF) | 0
  Res. Azithromycin (BALF): number analyzed (Participants) | 98
  Res. Azithromycin (BALF) | 14
  Sus. Azithromycin (NPS) | 106
  Int. Azithromycin (NPS) | 0
  Res. Azithromycin (NPS) | 4
  Sus. Tetracycline (BALF): number analyzed (Participants) | 98
  Sus. Tetracycline (BALF) | 98
  Int. Tetracycline (BALF): number analyzed (Participants) | 98
  Int. Tetracycline (BALF) | 0
  Res. Tetracycline (BALF): number analyzed (Participants) | 98
  Res. Tetracycline (BALF) | 0
  Sus. Tetracycline (NPS) | 110
  Int. Tetracycline (NPS) | 0
  Res. Tetracycline (NPS) | 0
  Sus. Levofloxacin (BALF): number analyzed (Participants) | 98
  Sus. Levofloxacin (BALF) | 98
  Int. Levofloxacin (BALF): number analyzed (Participants) | 98
  Int. Levofloxacin (BALF) | 0
  Res. Levofloxacin (BALF): number analyzed (Participants) | 98
  Res. Levofloxacin (BALF) | 0
  Sus. Levofloxacin (NPS) | 110
  Int. Levofloxacin (NPS) | 0
  Res. Levofloxacin (NPS) | 0
  Sus. Trimethoprim/Sulfamethoxazole (BALF): number analyzed (Participants) | 98
  Sus. Trimethoprim/Sulfamethoxazole (BALF) | 56
  Int. Trimethoprim/Sulfamethoxazole (BALF): number analyzed (Participants) | 98
  Int. Trimethoprim/Sulfamethoxazole (BALF) | 35
  Res. Trimethoprim/Sulfamethoxazole (BALF): number analyzed (Participants) | 98
  Res. Trimethoprim/Sulfamethoxazole (BALF) | 7
  Sus. Trimethoprim/Sulfamethoxazole (NPS) | 103
  Int. Trimethoprim/Sulfamethoxazole (NPS) | 7
  Res. Trimethoprim/Sulfamethoxazole(NPS) | 0

20. Secondary Outcome: Descriptive Statistics of the Antimicrobial Susceptibility Response of M. Catarrhalis for Unique Isolates Among Qualitative Positive Subjects, for Penicilin
Description: Antibiotic response of M. catarrhalis was tested against antibiotics which included: Penicilin.
  Samples assessed were BAL fluid (BALF) samples and Nasopharyngeal swab (NPS) samples.
  Unique isolate definition: 2 isolates of S.p., H.i. and M.c. were selected per specimen type per subjects. For analyses, the 2 isolates were compared to determine if they were clones vs. different ("unique") pathogen. Isolates were considered "unique" based on the comparison of serotype and antibiotic susceptibility (AS) profile for S.p. and H.i. and on the AS profile alone for M.c.. If the 2 isolates had different serotypes, or the same serotype but a different AS profile, then the 2 isolates were considered "unique", and both isolates were retained in the analyses.
  Note: For one subject who underwent BAL procedure, no BAL fluid was available for study analyses.
Time Frame: From Day 0 to Year 2
Population: as for outcome 19
Measure: Median (Full Range); unit: unique isolates of subjects
Arm/Group | Total Group
Number analyzed (Participants) | 110
unique isolates of subjects
  Penicilin (BALF): number analyzed (Participants) | 98
  Penicilin (BALF) | 8.00 [0.02 to 16.00]
  Penicilin (NPS) | 16.00 [0.02 to 16.00]

21. Secondary Outcome: Number of H. Influenzae or M. Catarrhalis Unique Isolates With Antimicrobial Susceptibility Positive Response Among Qualitative Positive Siubjects for Beta-lactamase
Description: Antimicrobial response of H. influenzae and M. catarrhalis was tested for Beta-lactamase (following Clinical and Laboratory Standards Institute [CLSI] guidelines [CLSI, 2015]).
  Samples assessed were BAL fluid (BALF) samples and Nasopharyngeal swab (NPS) samples.
  Unique isolate definition: 2 isolates of S.p., H.i. and M.c. were selected per specimen type per subjects. For analyses, the 2 isolates were compared to determine if they were clones vs. different ("unique") pathogen. Isolates were considered "unique" based on the comparison of serotype and antibiotic susceptibility (AS) profile for S.p. and H.i. and on the AS profile alone for M.c.. If the 2 isolates had different serotypes, or the same serotype but a different AS profile, then the 2 isolates were considered "unique", and both isolates were retained in the analyses.
  Note: For one subject who underwent BAL procedure, no BAL fluid was available for study analyses.
Time Frame: From Day 0 to Year 2
Population: The analysis was performed on the H. influenzae and M. catarrhalis unique isolates from qualitative positive subjects who were included in the ATP cohort.
Measure: Number; unit: unique isolates of subjects
Arm/Group | Total Group
Number analyzed (Participants) | 110
unique isolates of subjects
  H. influenzae (BALF): number analyzed (Participants) | 98
  H. influenzae (BALF) | 7
  H. influenzae (NPS): number analyzed (Participants) | 92
  H. influenzae (NPS) | 9
  M. catarrhalis (BALF): number analyzed (Participants) | 98
  M. catarrhalis (BALF) | 93
  M. catarrhalis (NPS) | 108

22. Secondary Outcome: Number of S. Pneumoniae Unique Isolates With Antimicrobial Susceptibility Response From Quantitative Positive Subjects
Description: as for outcome 16
Time Frame: From Day 0 to Year 2
Population: The analysis was performed on the S. pneumoniae unique isolates from quantitative positive subjects who were included in the ATP cohort.
Measure: Number; unit: Unique isolates of subjects
Arm/Group | Total Group
Number analyzed (Participants) | 26
Unique isolates of subjects
  Sus. Penicilin (BALF): number analyzed (Participants) | 21
  Sus. Penicilin (BALF) | 15
  Int. Penicilin (BALF): number analyzed (Participants) | 21
  Int. Penicilin (BALF) | 2
  Res. Penicilin (BALF): number analyzed (Participants) | 21
  Res. Penicilin (BALF) | 4
  Sus. Penicilin (NPS) | 11
  Int. Penicilin (NPS) | 10
  Res. Penicilin (NPS) | 5
  Sus. Amoxicillin/Clavulanate (BALF): number analyzed (Participants) | 21
  Sus. Amoxicillin/Clavulanate (BALF) | 17
  Int. Amoxicillin/Clavulanate (BALF): number analyzed (Participants) | 21
  Int. Amoxicillin/Clavulanate (BALF) | 3
  Res. Amoxicillin/Clavulanate (BALF): number analyzed (Participants) | 21
  Res. Amoxicillin/Clavulanate (BALF) | 1
  Sus. Amoxicillin/Clavulanate (NPS) | 22
  Int. Amoxicillin/Clavulanate (NPS) | 3
  Res. Amoxicillin/Clavulanate (NPS) | 1
  Sus. Erythromycin (BALF): number analyzed (Participants) | 21
  Sus. Erythromycin (BALF) | 17
  Int. Erythromycin (BALF): number analyzed (Participants) | 21
  Int. Erythromycin (BALF) | 0
  Res. Erythromycin (BALF): number analyzed (Participants) | 21
  Res. Erythromycin (BALF) | 4
  Sus. Erythromycin (NPS) | 11
  Int. Erythromycin (NPS) | 0
  Res. Erythromycin (NPS) | 15
  Sus. Azithromycin (BALF): number analyzed (Participants) | 21
  Sus. Azithromycin (BALF) | 15
  Int. Azithromycin (BALF): number analyzed (Participants) | 21
  Int. Azithromycin (BALF) | 2
  Res. Azithromycin (BALF): number analyzed (Participants) | 21
  Res. Azithromycin (BALF) | 4
  Sus. Azithromycin (NPS) | 11
  Int. Azithromycin (NPS) | 2
  Res. Azithromycin (NPS) | 13
  Sus. Tetracycline (BALF): number analyzed (Participants) | 21
  Sus. Tetracycline (BALF) | 18
  Int. Tetracycline (BALF): number analyzed (Participants) | 21
  Int. Tetracycline (BALF) | 0
  Res. Tetracycline (BALF): number analyzed (Participants) | 21
  Res. Tetracycline (BALF) | 3
  Sus. Tetracycline (NPS) | 16
  Int. Tetracycline (NPS) | 1
  Res. Tetracycline (NPS) | 9
  Sus. Levofloxacin (BALF): number analyzed (Participants) | 21
  Sus. Levofloxacin (BALF) | 21
  Int. Levofloxacin (BALF): number analyzed (Participants) | 21
  Int. Levofloxacin (BALF) | 0
  Res. Levofloxacin (BALF): number analyzed (Participants) | 21
  Res. Levofloxacin (BALF) | 0
  Sus. Levofloxacin (NPS) | 25
  Int. Levofloxacin (NPS) | 0
  Res. Levofloxacin (NPS) | 1
  Sus. Trimethoprim/Sulfamethoxazole (BALF): number analyzed (Participants) | 21
  Sus. Trimethoprim/Sulfamethoxazole (BALF) | 3
  Int. Trimethoprim/Sulfamethoxazole (BALF): number analyzed (Participants) | 21
  Int. Trimethoprim/Sulfamethoxazole (BALF) | 5
  Res. Trimethoprim/Sulfamethoxazole (BALF): number analyzed (Participants) | 21
  Res. Trimethoprim/Sulfamethoxazole (BALF) | 13
  Sus. Trimethoprim/Sulfamethoxazole (NPS) | 12
  Int. Trimethoprim/Sulfamethoxazole (NPS) | 2
  Res. Trimethoprim/Sulfamethoxazole (NPS) | 12

23. Secondary Outcome: Number of H. Influenzae Unique Isolates With Antimicrobial Susceptibility Response From Quantitative Positive Subjects
Description: Antibiotic response of H.ifluenzae was susceptible (Sus), or intermediate (Int), or resistant (Res)(following Clinical and Laboratory Standards Institute [CLSI] guidelines [CLSI, 2015])towards the tested antibiotics which included: Amoxicillin/Clavulanate, Azithromycin, Tetracycline, Levofloxacin, Trimethoprim/Sulfamethoxazole.
  Samples assessed were BAL fluid (BALF) samples and Nasopharyngeal swab (NPS) samples.
  For the "Unique isolate definition", please refer to the previous outcomes description.
  Note: For one subject who underwent BAL procedure, no BAL fluid was available for study analyses.
Time Frame: From Day 0 to Year 2
Population: The analysis was performed on the H. influenzae unique isolates from quantitative positive subjects who were included in the ATP cohort.
Measure: Number; unit: Unique isolates of subjects
Arm/Group | Total Group
Number analyzed (Participants) | 18
Unique isolates of subjects
  Sus. Amoxicillin/Clavulanate (BALF) | 15
  Int. Amoxicillin/Clavulanate (BALF) | 0
  Res. Amoxicillin/Clavulanate (BALF) | 3
  Sus. Amoxicillin/Clavulanate (NPS): number analyzed (Participants) | 8
  Sus. Amoxicillin/Clavulanate (NPS) | 8
  Int. Amoxicillin/Clavulanate (NPS): number analyzed (Participants) | 8
  Int. Amoxicillin/Clavulanate (NPS) | 0
  Res. Amoxicillin/Clavulanate (NPS): number analyzed (Participants) | 8
  Res. Amoxicillin/Clavulanate (NPS) | 0
  Sus. Azithromycin (BALF) | 17
  Int. Azithromycin (BALF) | 0
  Res. Azithromycin (BALF) | 1
  Sus. Azithromycin (NPS): number analyzed (Participants) | 8
  Sus. Azithromycin (NPS) | 8
  Int. Azithromycin (NPS): number analyzed (Participants) | 8
  Int. Azithromycin (NPS) | 0
  Res. Azithromycin (NPS): number analyzed (Participants) | 8
  Res. Azithromycin (NPS) | 0
  Sus. Tetracycline (BALF) | 18
  Int. Tetracycline (BALF) | 0
  Res. Tetracycline (BALF) | 0
  Sus. Tetracycline (NPS): number analyzed (Participants) | 8
  Sus. Tetracycline (NPS) | 8
  Int. Tetracycline (NPS): number analyzed (Participants) | 8
  Int. Tetracycline (NPS) | 0
  Res. Tetracycline (NPS): number analyzed (Participants) | 8
  Res. Tetracycline (NPS) | 0
  Sus. Levofloxacin (BALF) | 18
  Int. Levofloxacin (BALF) | 0
  Res. Levofloxacin (BALF) | 0
  Sus. Levofloxacin (NPS): number analyzed (Participants) | 8
  Sus. Levofloxacin (NPS) | 8
  Int. Levofloxacin (NPS): number analyzed (Participants) | 8
  Int. Levofloxacin (NPS) | 0
  Res. Levofloxacin (NPS): number analyzed (Participants) | 8
  Res. Levofloxacin (NPS) | 0
  Sus. Trimethoprim/Sulfamethoxazole (BALF) | 5
  Int. Trimethoprim/Sulfamethoxazole (BALF) | 7
  Res. Trimethoprim/Sulfamethoxazole (BALF) | 6
  Sus. Trimethoprim/Sulfamethoxazole (NPS): number analyzed (Participants) | 8
  Sus. Trimethoprim/Sulfamethoxazole (NPS) | 5
  Int. Trimethoprim/Sulfamethoxazole (NPS): number analyzed (Participants) | 8
  Int. Trimethoprim/Sulfamethoxazole (NPS) | 0
  Res. Trimethoprim/Sulfamethoxazole (NPS): number analyzed (Participants) | 8
  Res. Trimethoprim/Sulfamethoxazole (NPS) | 3

24. Secondary Outcome: Descriptive Statistics of the Antimicrobial Susceptibility Response of H.Influenzae for Unique Isolates Among Quantitative Positive Subjects, for Penicilin and Erythromycin
Description: Antibiotic response of H.ifluenzae was tested against antibiotics which included: Penicilin and Erythromycin (following Clinical and Laboratory Standards Institute [CLSI] guidelines [CLSI, 2015]).
  Samples assessed were BAL fluid (BALF) samples and Nasopharyngeal swab (NPS) samples.
  Unique isolate definition: 2 isolates of S.p., H.i. and M.c. were selected per specimen type per subjects. For analyses, the 2 isolates were compared to determine if they were clones vs. different ("unique") pathogen. Isolates were considered "unique" based on the comparison of serotype and antibiotic susceptibility (AS) profile for S.p. and H.i. and on the AS profile alone for M.c.. If the 2 isolates had different serotypes, or the same serotype but a different AS profile, then the 2 isolates were considered "unique", and both isolates were retained in the analyses.
  Note: For one subject who underwent BAL procedure, no BAL fluid was available for study analyses.
Time Frame: From Day 0 to Year 2
Population: as for outcome 23
Measure: Median (Full Range); unit: Unique isolates of subjects
Arm/Group | Total Group
Number analyzed (Participants) | 18
Unique isolates of subjects
  Penicilin (BALF) | 0.50 [0.25 to 16.00]
  Penicilin (NPS): number analyzed (Participants) | 8
  Penicilin (NPS) | 0.5 [0.13 to 16.00]
  Erythromycin (BALF) | 4.00 [2.00 to 16.00]
  Erythromycin (NPS): number analyzed (Participants) | 8
  Erythromycin (NPS) | 4.00 [2.00 to 8.00]

25. Secondary Outcome: Number of M. Catarrhalis Unique Isolates With Antimicrobial Susceptibility Response From Quantitative Positive Subjects
Description: Antibiotic response of M. catarrhalis was susceptible (Sus.), or intermediate (Int.), or resistant (Res.)(following Clinical and Laboratory Standards Institute [CLSI] guidelines [CLSI, 2015]) towards the tested antibiotics which included: Amoxicillin/Clavulanate, Erythromycin, Azithromycin, Tetracycline, Levofloxacin, Trimethoprim/Sulfamethoxazole.
  Samples assessed were BAL fluid (BALF) samples and Nasopharyngeal swab (NPS) samples.
  For the "Unique isolate definition", please refer to the previous outcome description.
  Note: For one subject who underwent BAL procedure, no BAL fluid was available for study analyses.
Time Frame: From Day 0 to Year 2
Population: The analysis was performed on the M. catarrhalis unique isolates from quantitative positive subjects who were included in the ATP cohort.
Measure: Number; unit: Unique isolates of subjects
Arm/Group | Total Group
Number analyzed (Participants) | 13
Unique isolates of subjects
  Sus. Amoxicillin/Clavulanate (BALF) | 12
  Int. Amoxicillin/Clavulanate (BALF) | 0
  Res. Amoxicillin/Clavulanate (BALF) | 1
  Sus. Amoxicillin/Clavulanate (NPS): number analyzed (Participants) | 10
  Sus. Amoxicillin/Clavulanate (NPS) | 9
  Int. Amoxicillin/Clavulanate (NPS): number analyzed (Participants) | 10
  Int. Amoxicillin/Clavulanate (NPS) | 0
  Res. Amoxicillin/Clavulanate (NPS): number analyzed (Participants) | 10
  Res. Amoxicillin/Clavulanate (NPS) | 1
  Sus. Erythromycin (BALF) | 12
  Int. Erythromycin (BALF) | 0
  Res. Erythromycin (BALF) | 1
  Sus. Erythromycin (NPS): number analyzed (Participants) | 10
  Sus. Erythromycin (NPS) | 9
  Int. Erythromycin (NPS): number analyzed (Participants) | 10
  Int. Erythromycin (NPS) | 0
  Res. Erythromycin (NPS): number analyzed (Participants) | 10
  Res. Erythromycin (NPS) | 1
  Sus. Azithromycin (BALF) | 11
  Int. Azithromycin (BALF) | 0
  Res. Azithromycin (BALF) | 2
  Sus. Azithromycin (NPS): number analyzed (Participants) | 10
  Sus. Azithromycin (NPS) | 9
  Int. Azithromycin (NPS): number analyzed (Participants) | 10
  Int. Azithromycin (NPS) | 0
  Res. Azithromycin (NPS): number analyzed (Participants) | 10
  Res. Azithromycin (NPS) | 1
  Sus. Tetracycline (BALF) | 13
  Int. Tetracycline (BALF) | 0
  Res. Tetracycline (BALF) | 0
  Sus. Tetracycline (NPS): number analyzed (Participants) | 10
  Sus. Tetracycline (NPS) | 10
  Int. Tetracycline (NPS): number analyzed (Participants) | 10
  Int. Tetracycline (NPS) | 0
  Res. Tetracycline (NPS: number analyzed (Participants) | 10
  Res. Tetracycline (NPS | 0
  Sus. Levofloxacin (BALF) | 13
  Int. Levofloxacin (BALF) | 0
  Res. Levofloxacin (BALF) | 0
  Sus. Levofloxacin (NPS): number analyzed (Participants) | 10
  Sus. Levofloxacin (NPS) | 10
  Int. Levofloxacin (NPS): number analyzed (Participants) | 10
  Int. Levofloxacin (NPS) | 0
  Res. Levofloxacin (NPS): number analyzed (Participants) | 10
  Res. Levofloxacin (NPS) | 0
  Sus. Trimethoprim/Sulfamethoxazole (BALF) | 7
  Int. Trimethoprim/Sulfamethoxazole (BALF) | 5
  Res. Trimethoprim/Sulfamethoxazole (BALF) | 1
  Sus. Trimethoprim/Sulfamethoxazole (NPS): number analyzed (Participants) | 10
  Sus. Trimethoprim/Sulfamethoxazole (NPS) | 10
  Int. Trimethoprim/Sulfamethoxazole (NPS): number analyzed (Participants) | 10
  Int. Trimethoprim/Sulfamethoxazole (NPS) | 0
  Res. Trimethoprim/Sulfamethoxazole (NPS): number analyzed (Participants) | 10
  Res. Trimethoprim/Sulfamethoxazole (NPS) | 0

26. Secondary Outcome: Descriptive Statistics of the Antimicrobial Susceptibility Response of M. Catarrhalis for Unique Isolates Among Quantitative Positive Subjects, for Penicilin
Description: Antibiotic response of M. catarrhalis was tested against antibiotics which included: Penicilin (following Clinical and Laboratory Standards Institute [CLSI] guidelines [CLSI, 2015]).
  Samples assessed were BAL fluid (BALF) samples and Nasopharyngeal swab (NPS) samples.
  Unique isolate definition: 2 isolates of S.p., H.i. and M.c. were selected per specimen type per subjects. For analyses, the 2 isolates were compared to determine if they were clones vs. different ("unique") pathogen. Isolates were considered "unique" based on the comparison of serotype and antibiotic susceptibility (AS) profile for S.p. and H.i. and on the AS profile alone for M.c.. If the 2 isolates had different serotypes, or the same serotype but a different AS profile, then the 2 isolates were considered "unique", and both isolates were retained in the analyses.
  Note: For one subject who underwent BAL procedure, no BAL fluid was available for study analyses.
Time Frame: From Day 0 to Year 2
Population: as for outcome 25
Measure: Median (Full Range); unit: Unique isolates of subjects
Arm/Group | Total Group
Number analyzed (Participants) | 13
Unique isolates of subjects
  Penicilin (BALF) | 16.00 [0.50 to 16.00]
  Penicilin (NPS): number analyzed (Participants) | 10
  Penicilin (NPS) | 16.00 [1.00 to 16.00]

27. Secondary Outcome: Number of H. Influenzae and M. Catarrhalis Unique Isolates With Antimicrobial Susceptibility Positive Response From Quantitative Positive Subjects, for Beta-lactamase
Description: as for outcome 21
Time Frame: From Day 0 to Year 2
Population: The analysis was performed on the H. influenzae or M. catarrhalis unique isolates from quantitative positive subjects who were included in the ATP cohort.
Measure: Number; unit: Unique isolates of subjects
Arm/Group | Total Group
Number analyzed (Participants) | 18
Unique isolates of subjects
  H. influenzae (BALF) | 3
  H. influenzae (NPS): number analyzed (Participants) | 8
  H. influenzae (NPS) | 1
  M. catarrhalis (BALF): number analyzed (Participants) | 13
  M. catarrhalis (BALF) | 13
  M. catarrhalis (NPS): number analyzed (Participants) | 10
  M. catarrhalis (NPS) | 10

28. Secondary Outcome: Mean Age of Subjects
Description: Demographic characteristics included age, which was expressed in months.
Time Frame: From Day 0 to Year 2
Population: The analysis was performed on the According to protocol (ATP) cohort, which included all evaluable subjects, who complied with the protocol and with BAL fluid sampling and/ or nasopharyngeal swab sampling results available.
Measure: Mean (Standard Deviation); unit: Months
Arm/Group | Total Group
Number analyzed (Participants) | 191
Months | 39.84 (17.76)

29. Secondary Outcome: Subject Gender
Description: Demographic characteristics included gender: female and male.
Time Frame: From Day 0 to Year 2
Population: as for outcome 28
Measure: Count of Participants; unit: Participants
Arm/Group | Total Group
Number analyzed (Participants) | 191
Participants
  Gender (Female) | 92
  Gender (Male) | 99

30. Secondary Outcome: Mean Weight of Subjects
Description: Demographic characteristics included weight which was expressed in kilograms (kg).
Time Frame: From Day 0 to Year 2
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | Total Group
Number analyzed (Participants) | 191
Kilograms | 14.67 (3.83)

31. Secondary Outcome: Mean Height of Subjects
Description: Demographic characteristics included height which was expressed in centimeters (cm).
Time Frame: From Day 0 to Year 2
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: Centimeters
Arm/Group | Total Group
Number analyzed (Participants) | 191
Centimeters | 96.04 (13.10)

32. Secondary Outcome: Number of Subjects With Body Mass Index (BMI) Characteristics
Description: Demographic characteristics included body mass index (BMI) whose z-scores were measures of relative weight adjusted for child age and sex.
Time Frame: From Day 0 to Year 2
Population: as for outcome 28
Measure: Count of Participants; unit: Participants
Arm/Group | Total Group
Number analyzed (Participants) | 191
Participants
  BMI - Marked thinness [< z-score (-3)] | 5
  BMI - Thinness [≥ z-score (-3) and < z-score (-2)] | 9
  BMI - Normal [≥ z-score (-2) and ≤ z-score (1)] | 122
  BMI - Overweight [> z-score (1) and ≤ z-score (2)] | 26
  BMI - Obesity [> z-score (2) and ≤ z-score (3)] | 14
  BMI - Extreme obesity [> z-score (3)] | 4

33. Secondary Outcome: Number of Subjects Presenting General Medical History Characteristics
Description: General medical history characteristics included: any pre-existing conditions, congenital chromosomal abnormality, prematurity (less than 37 weeks) neonatal problems, chronic renal failure, immune system disorder (including auto-immune), atopic dermatitis, clinician-confirmed eczema, asthma and other.
Time Frame: From Day 0 to Year 2
Population: as for outcome 28
Measure: Count of Participants; unit: Participants
Arm/Group | Total Group
Number analyzed (Participants) | 191
Participants
  Any other pre-existing conditions (Yes) | 176
  Any other pre-existing conditions (No) | 15
  Congenital chromosomal abnormality (Yes) | 2
  Prematurity (<37 weeks) (Yes) | 33
  Neonatal problems (Yes) | 18
  Chronic renal failure (Yes) | 1
  Immune system disorder (Yes) | 1
  History of inhaled steroids (Yes) | 134
  Atopic dermatitis (Yes) | 49
  Clinician-confirmed eczema (Yes) | 4
  Asthma (Yes) | 72
  Other (Yes) | 117

34. Secondary Outcome: Mean Gestational Age of Subjects
Description: General medical history included mean gestational age.
Time Frame: From Day 0 to Year 2
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: Weeks
Arm/Group | Total Group
Number analyzed (Participants) | 191
Weeks | 33.00 (2.95)

35. Secondary Outcome: Number of Subjects With Pneumococcal Vaccination History Characteristics
Description: Pneumococcal vaccination history characteristics included vaccination, pneumococcal vaccines received (Prevnar only, Prevnar 13 only, Synflorix only, Mix of vaccines), Prevnar only doses (1-4), Prevnar 13 only doses (1-4), Synflorix only doses (4), medical history source validated or not.
Time Frame: From Day 0 to Year 2
Population: as for outcome 28
Measure: Count of Participants; unit: Participants
Arm/Group | Total Group
Number analyzed (Participants) | 191
Participants
  Child has received any PCV (Yes) | 168
  Child has received only Prevenar | 15
  Child has received only Prevenar 13 | 123
  Child has received only Synflorix | 1
  Child has received Mix of vaccines | 29
  Doses of Prevenar (1) | 2
  Doses of Prevenar (2) | 4
  Doses of Prevenar (3) | 3
  Doses of Prevenar (4) | 6
  Doses of Prevenar 13 (1) | 4
  Doses of Prevenar 13 (2) | 12
  Doses of Prevenar 13 (3) | 46
  Doses of Prevenar 13 (4) | 61
  Doses of Synflorix (4) | 1
  Validated source | 165
  Not validated source | 3

36. Secondary Outcome: Number of Subjects With Flu Vaccination History Characteristics
Description: Flu vaccination history included vaccination, Flu vaccine doses (1-5), medical history source validated or not.
Time Frame: From Day 0 to Year 2
Population: as for outcome 28
Measure: Count of Participants; unit: Participants
Arm/Group | Total Group
Number analyzed (Participants) | 191
Participants
  Child has ever received any flu vaccine (Yes) | 58
  Number of doses of any flu vaccine (1) | 18
  Number of doses of any flu vaccine (2) | 26
  Number of doses of any flu vaccine (3) | 6
  Number of doses of any flu vaccine (4) | 5
  Number of doses of any flu vaccine (5) | 3
  Validated source | 52
  Not validated source | 6

37. Secondary Outcome: Number of Subjects With Haemophilus Influenzae Type b Vaccination History Characteristics
Description: Haemophilus influenzae type b vaccination history included vaccination, Haemophilus influenzae type b vaccine doses (1-4), medical history source validated or not.
Time Frame: From Day 0 to Year 2
Population: as for outcome 28
Measure: Count of Participants; unit: Participants
Arm/Group | Total Group
Number analyzed (Participants) | 191
Participants
  Child has received H.I. type b vaccine (Yes) | 188
  Number of doses of H.I. type b vaccine (1) | 2
  Number of doses of H.I. type b vaccine (2) | 4
  Number of doses of H.I. type b vaccine (3) | 38
  Number of doses of H.I. type b vaccine (4) | 144
  Validated source | 184
  Not validated source | 4

38. Secondary Outcome: Number of Subjects With Antibiotics and Other Medications Administered
Description: Medication history referred to antibiotics administered in the past 6 months, drug names, antibiotic information source, other medications administered during the past 6 months, information source.
Time Frame: From Day 0 to Year 2
Population: as for outcome 28
Measure: Count of Participants; unit: Participants
Arm/Group | Total Group
Number analyzed (Participants) | 191
Participants
  Antibiotic administered in the past 6 months (Yes) | 153
  Penicillin | 83
  Amoxicillin/ Clavulanate | 76
  Cephalosporins | 24
  Erythromycin | 1
  Azithromycin | 57
  Clarithromycin | 8
  Ciprofloxacin | 2
  Clindamycin | 1
  Linezolid | 1
  Meropenem | 1
  Antibiotics source information. - parent recall | 49
  Antibiotics source information. - medical file | 120
  Other medications in the past 6 months (Yes) | 177
  Source of information. - parent recall | 49
  Source of information. - medical file | 149

39. Secondary Outcome: Number of Subjects With Clinical Characteristics
Description: Clinical characteristics included affections/pre-conditions, affection episodes, number of children living in a household, children in day-care centres, exposure to cigarette smoke.
Time Frame: From Day 0 to Year 2
Population: as for outcome 28
Measure: Count of Participants; unit: Participants
Arm/Group | Total Group
Number analyzed (Participants) | 191
Participants
  Cough (Yes) | 151
  Wheezing (Yes) | 86
  Pathologic auscultation (Yes) | 74
  Infiltrates atelectasis diagnosed by X-ray (Yes) | 131
  Wet cough lasting 4 weeks without additional (Yes) | 63
  Persistent wheezing lasting 3 months (Yes) | 8
  Recurrent wheezing 3 or more episodes/year (Yes) | 25
  Persistent pathologic auscultation (Yes) | 16
  Persistent 1 month infiltrates atelectasis (Yes) | 65
  3 episodes/year infiltrates atelectasis (Yes) | 14
  Any respiratory/otitis media pre-conditions(Yes) | 186
  Any respiratory/otitis media pre- conditions (No) | 5
  Pneumonia (Yes) | 114
  Bronchiolitis (Yes) | 85
  Bronchioectasis (Yes) | 15
  Bronchitis (Yes) | 143
  Rhinitis (Yes) | 15
  Acute otitis media (Yes) | 53
  Otitis media with effusion or glue ear (Yes) | 6
  Otitis media with perforation and discharge (Yes) | 8
  The child had ever been breastfed (Yes) | 150
  The child had ever been breastfed (No) | 41
  The child was currently breastfed (Yes) | 6
  The child was currently breastfed (No) | 144
  Other children <6 years in the same household (0) | 101
  children <6 years in the same household (1-2) | 87
  children <6 years in the same household (≥3) | 3
  children ≥ 6 years in the same household (0) | 134
  children ≥ 6 years in the same household (1-2) | 55
  children ≥ 6 years in the same household (≥3) | 2
  Child at daycare &/school at least 2 day/week(Yes) | 155
  Child at day care &/school at least 2 day/week(No) | 36
  Child lived within 1 km of major polluters (Yes) | 63
  Child lived within 1 km of major polluters (No) | 128
  Major roadway (Yes) | 20
  Highway (Yes) | 27
  Area where trucks or vehicles were idle (Yes) | 11
  Major industry area with smokestacks (Yes) | 13
  Other (Yes) | 6
  Child with>3 day/week to cigarette smoke(Yes) | 38
  Child with>3 day/ week to cigarette smoked (No) | 153
  Previous episodes within the last year (0) | 2
  Previous episodes within the last year (1) | 11
  Previous episodes within the last year (2-3) | 52
  Previous episodes within the last year (4-5) | 45
  Previous episodes within the last year (6 or more) | 73
  Cough productive or wet (Yes) | 153
  Cough paroxysmal (Yes) | 29
  Cough laryngeal (Yes) | 38
  Shortness of breath independent of coughing (Yes) | 35
  Shortness of breath secondary to cough (Yes) | 33

40. Secondary Outcome: Number of Subjects With Laboratory Results
Description: Laboratory results included blood sample results available, white blood Cell (WBC) count analysed, WBC reference range, Clinically relevant to the suspected chronic lower respiratory tract infection (LRTI) in the child if out of the range of WBC [LRTI-WBC], CRP (C-reactive protein) reference range, CRP groups, Clinically relevant to the suspected chronic LRTI in the child if out of the range of CRP [LRTI-CRP], ESR (Erythrocyte sedimentation rate) analysed, ESR reference range and Clinically relevant to the suspected chronic LRTI in the child if out of the range of ESR [LRTI-ESR].
Time Frame: From Day 0 to Year 2
Population: as for outcome 28
Measure: Count of Participants; unit: Participants
Arm/Group | Total Group
Number analyzed (Participants) | 191
Participants
  Blood sample results available (Yes) | 109
  WBC count analysed (Yes) | 109
  WBC reference range (low-high ranges) | 78
  WBC reference range (>high range) | 31
  LRTI-WBC (Yes) | 18
  LRTI-WBC (No) | 17
  CRP analysed (Yes) | 57
  CRP analysed (No) | 52
  CRP reference range (low-high ranges) | 26
  CRP reference range (>high range) | 31
  CRP reference range (missing range) | 52
  CRP groups <40 mg/L | 46
  CRP groups ≥40-80 mg/L | 6
  CRP groups ≥80-120 mg/L | 3
  CRP groups ≥120 mg/L | 2
  LRTI-CRP (Yes) | 17
  LRTI-CRP (No) | 17
  ESR analysed (Yes) | 12
  ESR analysed (No) | 97
  ESR reference range (low-high ranges) | 8
  ESR reference range (>high range) | 4
  ESR reference range (missing range) | 97
  LRTI-ESR (Yes) | 2
  LRTI-ESR (No) | 3

41. Secondary Outcome: White Blood Cells (WBC) Laboratory Results
Description: Laboratory results for WBC were expressed in 10^9 cells per liter (10^9 cells/L).
Time Frame: From Day 0 to Year 2
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Total Group
Number analyzed (Participants) | 191
10^9 cells/L | 540.17 (2651.17)

42. Secondary Outcome: C-reactive Protein (CRP) Laboratory Results
Description: Laboratory results for CRP were expressed in milligrams per litre (mg/L).
Time Frame: From Day 0 to Year 2
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Total Group
Number analyzed (Participants) | 191
mg/L | 25.45 (37.91)

43. Secondary Outcome: Erythrocyte Sedimentation Rate (ESR) Laboratory Results
Description: Laboratory results for ESR were expressed in millimeters per hour (mm/hr).
Time Frame: From Day 0 to Year 2
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: mm/hr
Arm/Group | Total Group
Number analyzed (Participants) | 191
mm/hr | 25.33 (30.67)

44. Secondary Outcome: Number of Subjects With Radiological Results
Description: Radiological results included x-ray, result normality, relationship of abnormality to BAL sampling.
Time Frame: From Day 0 to Year 2
Population: as for outcome 28
Measure: Count of Participants; unit: Participants
Arm/Group | Total Group
Number analyzed (Participants) | 191
Participants
  A Chest X-ray was done (Yes) | 166
  A Chest X-ray was done (No) | 25
  Result (Normal) | 23
  Result (Abnormal) | 143
  Abnormality relevant to collecting the BALF(Yes) | 122
  Abnormality relevant to collecting the BALF (No) | 21

ADVERSE EVENTS:
Time Frame: SAE(s) considered related to the nasopharyngeal sampling procedure were reported during the entire study period, which lasted 2 years.
Description: No other (not including serious) adverse events were collected for this study, leading to 0 participants at risk in the Other adverse events section.
Arm/Group | Total Group
All-Cause Mortality (participants affected / at risk) | 0/197
Serious Adverse Events (participants affected / at risk) | 0/197
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2015-10-05): https://cdn.clinicaltrials.gov/large-docs/07/NCT02838407/Prot_000.pdf
  • Statistical Analysis Plan (2015-11-27): https://cdn.clinicaltrials.gov/large-docs/07/NCT02838407/SAP_001.pdf